CLINICAL TRIAL: NCT00741416
Title: Collection and Storage of Human Biological Materials (Blood Sample) and Linked Phenotypic Information (Health History) for Research Purposes
Brief Title: Biorepository: Indiana Health Study
Acronym: IHS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fairbanks Institute (Other)
Collaborators: Indiana University School of Medicine (Other); Richard M. Fairbanks Foundation (Other); BioCrossroads (Other); Regenstrief Institute, Inc. (Other)
Responsible Party: Cynthia J. Helphingstine, Fairbanks Institute for Healthy Communities
Other Study IDs: FI-08-US-0001
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Coronary Artery Disease; Heart Disease; Healthy
Keywords: Heart Disease; Biorepository; Biobank
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 70ml of whole blood: 3-10 ml EDTA tubes for collection of whole blood 3-10 ml SST tubes (red tops) for collection of serum 2-3ml PAXgene tubes for collection of RNA A minimum of 1 EDTA and 1 SST tube is required for enrollment into the study.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case: Those with a diagnosis of Coronary Artery Disease
- Control: Those who do not have Coronary Artery Disease (are healthy) but are matched to a Case participant by age, gender, and ethnicity.

SUMMARY:
Blood samples and health information (e.g., age at diagnosis, test results) are collected for the purposes of genetic research. The blood samples are assigned a number and stored in a repository for safe keeping until they are needed for a research project. Participants are persons who are healthy (not having high blood pressure, diabetes, or high cholesterol levels) or persons who have Coronary Artery Disease (CAD) and live in Indiana. Participants complete a questionnaire at the time the blood sample is drawn and are contacted once a year to update their health history. Researchers apply to the Fairbanks Institute for use of the blood samples and health information minus participant names and contact information. Their research is required to be related to find genes or substances made by genes that may be involved in Coronary Artery Disease with the purpose of improving the investigators understanding of the illness potentially leading to the development of new diagnostic tools for identifying the illness, new treatments,or preventative measures. This study will be repeated for other disorders like Diabetes and Cancer.

DETAILED DESCRIPTION:
Study Aim:

The purpose of this study is to create an extensively annotated bio-repository platform for hypothesis-driven research that will lead to advancements in the diagnosis, treatment and prevention of diseases common to the population of Indiana. The first phase of this research platform will be created by collecting blood samples from two groups of individuals in the Central Indiana community, one with documented evidence of coronary artery disease (CAD), and a second group of age, gender and ethnicity matched individuals without clinical evidence of CAD. Each individual's blood sample will be linked to their clinical, demographic and epidemiological information, gathered both retrospectively and prospectively. This will be repeated with individuals who have Cancer, Diabetes and potentially other illnesses.

Recruitment:

This initial study will include 750 individuals with CAD (the CAD Group) and 750 individuals who are age, gender, and ethnicity matched to the CAD Group, but without presentation of clinical evidence of CAD (the Control Group). To reflect the growing representation of Hispanics in Central Indiana, Hispanics will be overly recruited in both groups so that the study population accurately reflects the general population of Central Indiana.

Follow-up:

As this is a prospective, longitudinal study, follow-up of study subjects is intended to continue indefinitely, unless, of course, at any time, consent for further follow-up is withdrawn by the subject. Follow-up will include continuing access to the subject's medical record, as well as facilitating continued contact by telephone, to pursue data concerning changes in the subject's health. Subjects may be contacted by telephone, mail or email every twelve months to ask if they wish to continue participation in the study.

The collected dataset (made up of the collected blood samples linked to clinical and epidemiological information collected retrospectively and prospectively), will be used in medical research to find genes, or gene products such as RNA or proteins that will help in understanding the causes of disease and will guide the development of new treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Study subjects will be recruited for the CAD group based on a history confirmed by the medical record of at least one of the following:

* Angioplasty, with or without stent placement
* Coronary Artery Bypass Graft (CABG) surgery
* Diagnostic angiogram or positive catheterization results showing 50% occlusion or greater

Exclusion Criteria:

1. Study subjects for the Control Group will be excluded based on a confirmed history of:

   * CAD as defined above, or as history of a positive stress test for ischemia, Troponin > 0.5 or myocardial infarction
   * Diabetes (type 1 or 2)
   * Hypertension (confirmed with at least two documented measurements of blood pressure greater than 140/90, not attributed to treating medications)
   * Abnormal lipid profile defined as LDL-C < 130mg/dl, HDL ≥ 40 mg/dl, cholesterol < 240 mg/dl or triglycerides < 200 mg/dl
   * Patients taking any medications commonly used for the above excluded conditions
   * History of stroke or Transient Ischemic Attacks (TIAs)
2. Exclusion criteria for both the CAD Group and the Control Group will be a known or reported history of:

   * Hepatitis B
   * Hepatitis C
   * AIDS (HIV positive)
   * Tuberculosis
   * Cancer (including melanoma, but excluding low-malignancy skin cancer)
   * Non-autologous bone marrow transplant
   * Blood transfusion within 120 days
3. In addition, prisoners, minors, patients requiring the consent of a caregiver or Authorized Representative, and/or any subjects deemed medically unsuitable for research donation by their treating physician (for reasons such as anemia, hematopoetic disorders/cancers or low body weight) will be excluded from the study.
4. Subjects unwilling to consent to the allowance of future follow-up will be excluded from initial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This initial study will include 750 individuals with CAD (the CAD Group) and 750 individuals who are age, gender, and ethnicity matched to the CAD Group, but without presentation of clinical evidence of CAD (the Control Group). To reflect the growing representation of Hispanics in Central Indiana, Hispanics will be overly recruited in both groups so that the study population accurately reflects the general population of Central Indiana.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2008-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anantha Shekhar, MD PhD, Principal Investigator — Indiana University School of Medicine/CTSI; Cynthia Helphingstine, PhD, Study Director — Fairbanks Institute for Healthy Communities
Locations (14):
- United States (14):
  - American Health Network, Avon, Indiana
  - Investigator's Research Group, Brownsburg, Indiana
  - American Health Network, Franklin, Indiana
  - American Health Network, Greenfield, Indiana
  - Krannert Institute of Cardiology/IU Dept. of Medicine, Indianapolis, Indiana
  - Outpatient Clinical Research Facility/Indiana Cancer Pavilion, Indianapolis, Indiana
  - Indiana Heart Hospital: Community Heart and Vascular Clinic, Indianapolis, Indiana
  - Alivio Medical Center (spanish/espaniol), Indianapolis, Indiana
  - American Health Network, Indianapolis, Indiana
  - Oral Health Research Institute, Indianapolis, Indiana
  - Corvasc MDs, Indianapolis (North), Indiana
  - Indiana Heart Physicians, Indianapolis (South), Indiana
  - IU Health Arnett, Lafayette, Indiana
  - Medical Consultants, PC, Muncie, Indiana

REFERENCES:
- See also: Information on The Fairbanks Institute for Health Communities — http://www.fairbanksinstitute.org